CLINICAL TRIAL: NCT04122911
Title: A Phase II Single Arm Trial Evaluating the Efficacy and Safety of Temozolomide for Second-Line Treatment of Neuroendocrine Carcinomas Progressing After First-Line Platinum- Based Therapy
Brief Title: Temozolomide for Second-Line Treatment of Neuroendocrine Carcinomas
Acronym: TENEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TENEC
Record Dates: First submitted 2019-09-04; First posted 2019-10-10 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Neuroendocrine Carcinomas
Keywords: Temozolomide; second-line chemotherapy
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Temozolomide (Experimental): Temozolomide 75mg/m2 metronomic schedule: one week on/one week off in a cycle of 28 days
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — pharmacological

SUMMARY:
To assess the efficacy and safety of Temozolomide for second-line treatment of Neuroendocrine Carcinomas progressing after first-line Platinum-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-specific procedures or treatment, as confirmation of the patient's awareness and willingness to comply with the study requirements.
* Patients ≥18 years of age.
* Histologically confirmed Metastatic Neuroendocrine Carcinoma (Ki67>20% Ki67 must be quantified in percentage) with documented progression of disease per investigator assessment following or during first-line platinum-based treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2.
* At least 28 days since prior radiation therapy or surgery and recovery from treatment.
* Patients must have measurable disease which must be evaluable per RECIST v1.1.
* Estimated life expectancy of ≥12 weeks.

Exclusion Criteria:

* - Patients < 18 years of age
* Diagnosis of well differentiated G1/G2 NEN
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would prevent the patient from meeting the study requirements.
* Serious active infection requiring i.v. antibiotics and/or hospitalization at study entry.
* Patients who are treated with any medicinal product that contraindicates the use of the study drug, may interfere with the planned treatment, affects patient compliance or puts the patient at high risk for treatment-related complications.
* Pregnant or lactating females. Serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days with a confirmatory urine pregnancy test within 7 days prior to study treatment start. Women of childbearing potential (defined as <2 years after last menstruation and not surgically sterile) not using effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Patients with meningeal carcinomatosis
* Patients with organ allografts requiring immunosuppression
* Patients with known positive HIV status
* Patients with a hypersensitivity to Temozolomide or Dacarbazine
* Any laboratory values at baseline as follows:

Hematology:

1. Absolute Neutrophil Count (ANC) <1.5x109/L or 1500/mm3
2. Platelet count <100x109/L
3. Hemoglobin <8 g/dL (Note: hemoglobin levels may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors).

Coagulation:

1. International Normalized Ratio (INR) >1.5 except for patients on stable anticoagulant therapy
2. Activated Partial Thromboplastin Time (aPTT) ≥1.5 times upper limit of normal (ULN) or greater than the lower limit of the therapeutic range Note: The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least two weeks at the time of Day 1, Cycle 1.

Serum chemistry:

1. Total bilirubin >1.5 times ULN
2. Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) >2 times ULN (>5 times ULN for patients with known liver involvement)
3. Alkaline Phosphatase (ALP) >2 times ULN (>5 times ULN for patients with known liver involvement and >7 times ULN for patients with known bone involvement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01-29 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 months
  Overall response rate (ORR)

SECONDARY OUTCOMES:
Second Line Progression Free Survival (PFS) | 12 months
  Second Line Progression Free Survival (PFS)
Overall survival (OS) | 12 months
  Overall survival (OS)
Clinical Benefit Rate (CBR) | 12 month
  Clinical benefit rate (CBR) was defined as the proportion of patients with a complete or partial response or with stable disease (Complete Response + Partial Response + Stable Disease [CR+PR+SD]) at Week 24.
Safety and tolerability - Incidence of treatment-related adverse events (AE). | 1 month
  The NCI-CTCAE version 4.0 will be used to evaluate the clinical safety of the treatment in this study. Intensity of all adverse events (AEs) will be graded according to the NCI-CTCAE v 4.0 on a five-point scale (Grade 1 to 5). AEs not listed on the NCI-CTCAE should be graded according below. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life threatening/disabling; Grade 5: Death.
Safety and tolerability - Incidence of abnormal laboratory test results | 1 month
  The following assessments will be conducted in order to monitor patient safety:
  1. Hematology tests as per institutional standards.
  2. Biochemistry tests as per institutional standards.
  3. Coagulation tests as per institutional standards.
  4. Pregnancy test for women of child-bearing potential.
Safety and tolerability - Incidence of abnormal vital signs | 1 month
  * Blood pressure (mm/Hg)
  * Temperature (°C)
Safety and tolerability - Incidence of abnormal ECG readings | 1 month
  This examination is essential to highlight the presence of:
  * arrhythmias,
  * discontinuous heart rhythm changes,
  * ischemia, i.e. reduced blood supply to the heart,
  * presence of ailments such as heartbeat, chest pain, loss of consciousness or dizziness.
Quality of Life (QoL) - QoL will be assessed using the European Organization for Research and Trial in Cancer QOL core (EORTC QLQ-C30) questionnaire (version 3) [Quality of life questionnaire - QLQ] | 1 month
  The EORTC QLQ-C30 is a questionaire of 30-item and it incorporates 9 multi-item scales:5 functional scales (Physical,Role,Cognitive,Emotional and Social Functioning);3 symptom scales (Fatigue,Pain and Nausea/Vomiting) and a Global Health Status/QoL scale.6 single item scales are also included (Dyspnoea,Insomnia,Appetite Loss,Constipation,Diarrhoea and Financial Difficulties).Version 3.0 has 4-point scales for the first 5 items comprising the Physical Functioning scale.These are coded with the same response categories as items 6 to 28,namely "1 Not at all" (minimum value),"2 A little","3 Quite a bit" and "4 Very much" (maximum value).The last 2 question foresee a 7-point response scale:minimum value is "1 Very poor",maximum value is "7 Excellent".
Quality of Life (QoL) - QoL will be assessed using disease specific modules for Neuroendocrine Tumors (NET), the EORTC QLQ GINET21 (EORTC QLQ Gastrointestinal Neuroendocrine Tumors 21). | 1 month
  The QLQ-GINET21 contains 21 items:4 single-item assessments relating to muscle and/or bone pain (MBP),body image (BI),information (INF) and sexual functioning (SX),together with 17 items organised into 5 proposed scales:endocrine symptoms (ED 3 items),GI symptoms (GI 5 items),treatment-related symptoms (TR 3 items),social functioning (SF) of the new module (SF21, 3 items) and disease-related worries (DRW 3 items).The response format of the questionnaire is a 4-point Likert scale:"1 Not at all" (minimum value),"2 A little","3 Quite a bit" and "4 Very much" (maximum value).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Tumori di Napoli - Fondazione G. Pascale, Napoli, Campania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Arx C, Della Vittoria Scarpati G, Cannella L, Clemente O, Marretta AL, Bracigliano A, Picozzi F, Iervolino D, Granata V, Modica R, Bianco A, Mocerino C, Di Mauro A, Pizzolorusso A, Di Sarno A, Ottaiano A, Tafuto S; ENETs Center of Excellence in Naples, Italy and with the endorsement of the Italian Association for Neuroendocrine Tumor IT.A.NET. A new schedule of one week on/one week off temozolomide as second-line treatment of advanced neuroendocrine carcinomas (TENEC-TRIAL): a multicenter, open-label, single-arm, phase II trial. ESMO Open. 2024 May;9(5):103003. doi: 10.1016/j.esmoop.2024.103003. Epub 2024 Apr 13. PMID 38615472